CLINICAL TRIAL: NCT00988013
Title: A Phase I Study of Intensity Modulated Total Marrow Irradiation (IM-TMI) in Addition to Fludarabine/Busulfan Conditioning for Allogeneic Transplantation for Advanced Hematologic Malignancies
Brief Title: Intensity Modulated Total Marrow Irradiation (IM-TMI) for Advanced Hematologic Malignancies
Acronym: IM-TMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Damiano Rondelli, MD, Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0251
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; Lymphoblastic Leukemia; Acute Leukemia; Non Hodgkins Lymphoma; Chronic Myeloid Leukemia
Keywords: total marrow irradiation; intensity modulated radiation; leukemia; hematologic diseases
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: Dose escalation of total marrow irradiation prior to stem cell transplantation
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IM-TMI (3Gy) (Experimental): Patients will receive 3Gy per day for 1 day (total of 3Gy).
  Interventions: Radiation: IM-TMI (3Gy)
- IM-TMI (6Gy) (Experimental): Patients will receive 3Gy per day for 2 days (for a total of 6Gy).
  Interventions: Radiation: IM-TMI (6Gy)
- IM-TMI (9Gy) (Experimental): Patients will receive 3Gy per day for 3 days (for a total of 9Gy).
  Interventions: Radiation: IM-TMI (9Gy)
- IM-TMI (12Gy) (Experimental): Patients will receive 3Gy per day for 4 days (for a total of 12Gy).
  Interventions: Radiation: IM-TMI (12Gy)

INTERVENTIONS:
Radiation: IM-TMI (3Gy) — Patients will receive 3Gy per day for 1 day.
  Arms: IM-TMI (3Gy)
Radiation: IM-TMI (6Gy) — Patients will receive 3Gy per day for 2 days.
  Arms: IM-TMI (6Gy)
Radiation: IM-TMI (9Gy) — Patients will receive 3Gy per day for 3 days.
  Arms: IM-TMI (9Gy)
Radiation: IM-TMI (12Gy) — Patients will receive 3Gy per day for 4 days.
  Arms: IM-TMI (12Gy)

SUMMARY:
This is a phase I study using Intensity Modulated Total Marrow Irradiation (IM-TMI) in addition to a chemotherapy regimen in preparation for an allogeneic stem cell transplant for advanced hematologic malignancies such as acute myeloid or lymphoblastic leukemia, high grade non Hodgkin's or Hodgkin's lymphoma, chronic myelogenous leukemia, and plasma cell leukemia. Because the subjects participating in this study have a disease that is severe and has a high risk of relapse even after transplant, the investigators propose to use a chemotherapy regimen (fludarabine/busulfan), the name for the combination of chemotherapy drugs that is given to patients prior to transplantation of the donor stem cells, along with intensity modulated radiation (IM-TMI) to the bone marrow. Total body irradiation (TBI) in conjunction with chemotherapy is a standard of care as a pre-conditioning regimen prior to bone marrow transplant (BMT) in patients with hematologic malignancies. However, TBI can cause severe side effects due to irradiation of organs such as the lenses of the eye, whole brain, lungs, liver, kidneys, heart, small bowel and oral cavity. IM-TMI allows for the delivery of adequate doses of radiation to the bone marrow while sparing other organs and therefore limiting radiation side effects. The irradiation, along with receiving the chemotherapy drugs will suppress the subject's immune system and kill off tumor cells, but will also intensify the effect of the conditioning regimen thus allowing the bone marrow transplantation to have a greater chance of being successful.

No investigational drugs are used in this study. The investigational part of this study is the use of intensity modulated total marrow irradiation instead of conventional radiation. IMTMI can deliver 99% of the prescribed treatment to the targeted bones and reduce the doses of radiation to surrounding organs, as received in conventional TBI, by 29% to 65%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following diseases:

  * Acute myeloid or lymphoblastic leukemia in first complete remission if poor prognosis documented by failure to response after initial induction chemotherapy, or cytogenetic, or molecular studies.
  * Acute leukemia in greater/equal second remission, or partial remission after chemotherapy.
  * High grade non Hodgkin's or Hodgkin's lymphoma with marrow involvement resistant/ relapsed after second line therapy including high dose chemotherapy and autologous SCT.
  * CML in advanced or blastic phase.
  * Plasma cell leukemia.
* Age 18-60 years.
* Karnofsky performance status of 70
* Adequate cardiac and pulmonary function. Patients with decreased LVEF less than/equal to 40% or DLCO less than/equal to 50% of predicted will require clearance from cardiology or pulmonary services, respectively, prior to enrollment on this protocol.
* Serum creatinine less than/equal to 1.5 mg/dL or Creatinine Clearance greater than/equal to 50 ml/min .
* Serum bilirubin 2.0 mg/dl, SGPT less than/equal to 3 times the upper limit of normal

Exclusion Criteria:

* Life expectancy is severely limited by concomitant illness.
* Evidence of chronic active hepatitis or cirrhosis
* HIV-positive
* Patient is pregnant
* Patient or guardian is not able to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2009-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Rondelli, MD, Study Chair — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patel P, Aydogan B, Koshy M, Mahmud D, Oh A, Saraf SL, Quigley JG, Khan I, Sweiss K, Mahmud N, Peace DJ, DeMasi V, Awan AM, Weichselbaum RR, Rondelli D. Combination of linear accelerator-based intensity-modulated total marrow irradiation and myeloablative fludarabine/busulfan: a phase I study. Biol Blood Marrow Transplant. 2014 Dec;20(12):2034-41. doi: 10.1016/j.bbmt.2014.09.005. Epub 2014 Sep 16. PMID 25234438

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IM-TMI (3Gy) | IM-TMI (6Gy) | IM-TMI (9Gy) | IM-TMI (12Gy)
Started | 3 | 3 | 6 | 2
Completed | 3 | 3 | 6 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IM-TMI (3Gy) | IM-TMI (6Gy) | IM-TMI (9Gy) | IM-TMI (12Gy) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 2 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6 | 2 | 14
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 52 [52 to 63] | 38 [38 to 52] | 39 [20 to 65] | 53 [53 to 62] | 52 [20 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 7
  Male | 1 | 1 | 4 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 1 | 6
  Not Hispanic or Latino | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 3 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 3 | 2 | 4 | 2 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 | 2 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 4 TMI Toxicity
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Groups:
- IM-TMI (12Gy): Patients will receive 3Gy per day for 3 days (for a total of 12Gy).
  IM-TMI (9Gy): Patients will receive 3Gy per day for 3 days.
- IM-TMI (9Gy): Patients will receive 3Gy per day for 4 days (for a total of 9Gy).
  IM-TMI (12Gy): Patients will receive 3Gy per day for 4 days.
Arm/Group | IM-TMI (3Gy) | IM-TMI (6Gy) | IM-TMI (12Gy) | IM-TMI (9Gy)
Number analyzed (Participants) | 3 | 3 | 6 | 2
Participants | 0 | 0 | 0 | 2

2. Secondary Outcome: Time to Neutrophil and Platelet Engraftment in Patients With Hematologic Malignancies
Time Frame: Up to 100 days post-transplant
Measure: Median (Full Range); unit: Days
Arm/Group | IM-TMI (3Gy) | IM-TMI (6Gy) | IM-TMI (9Gy) | IM-TMI (12Gy)
Number analyzed (Participants) | 3 | 3 | 6 | 2
Days | 15 [10 to 20] | 15 [10 to 20] | 15 [10 to 20] | 15 [10 to 20]

3. Primary Outcome: Number of Participants With 1 Year Mortality Unrelated to TMI
Time Frame: 1 year post-transplant
Population: Grade 4 TMI toxicity 0 Grade 4 TMI toxicity 0 Grade 4 TMI toxicity 0 Grade 4 TMI toxicity 0
Measure: Count of Participants; unit: Participants
Arm/Group | IM-TMI (3Gy) | IM-TMI (6Gy) | IM-TMI (9Gy) | IM-TMI (12Gy)
Number analyzed (Participants) | 3 | 3 | 6 | 2
Participants | 0 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | IM-TMI (3Gy) | IM-TMI (6Gy) | IM-TMI (9Gy) | IM-TMI (12Gy)
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 4/6 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 2/6 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM-TMI (3Gy) (N=3) | IM-TMI (6Gy) (N=3) | IM-TMI (9Gy) (N=6) | IM-TMI (12Gy) (N=2)
GI hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GVHD (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IM-TMI (3Gy) (N=3) | IM-TMI (6Gy) (N=3) | IM-TMI (9Gy) (N=6) | IM-TMI (12Gy) (N=2)
Oral mucositis (Infections and infestations) | 3 (3) | 3 (3) | 6 (6) | 2 (2)
Gut mucocitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No